CLINICAL TRIAL: NCT00329069
Title: Vascular Endothelial Receptor Activity in Patients With Coronary Artery Disease on Medication With Statins
Brief Title: The Role of Atorvastatin on Monocyte Function in Patients With Coronary Artery Disease and Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ATV-D-01-007 G
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2006-05-24 (Estimated); Status verified 2006-05

CONDITIONS: Coronary Artery Disease; Hypercholesterolemia; Monocyte Function
Keywords: statin; atorvastatin; hypercholesterolemia; coronary artery disease; monocyte; collateral formation; arteriogenesis; chemotaxis; migration; growth factors; vascular endothelial growth factor A; placenta growth factor 1; hepatocyte growth factor; monocyte chemotactic protein 1
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia; Chemotaxis; Deafness, Autosomal Recessive 39 | interventions — Atorvastatin; Pharmaceutical Preparations

INTERVENTIONS:
Drug: atorvastatin (drug)

SUMMARY:
The aim of this study is to determine, whether an intensified atorvastatin therapy can improve monocyte function in patients with coronary artery disease and hypercholesterolemia.

DETAILED DESCRIPTION:
Hypercholesterolemia is one of the most important cardiovascular risk factors that significantly elevates the risk for the development and progression of arteriosclerotic diseases.

Statins such as atorvastatin have been shown to reduce atherogenic lipoprotein levels as well as cardiovascular morbidity and mortality in a large number of clinical trials. It is suggested that statins have- apart from their lipid-lowering properties- other pleiotropic effects that are responsible for their anti-atheroslerotic and and cardioprotective potential.

Monocytes are crucially involved in the process of arteriogenesis (i.e. the growth of preexisting arterioles). Monocyte chemotaxis can be stimulated with arteriogenic molecules such as vascular endothelial growth factor A (VEGF-A). In previous studies we could demonstrate that the VEGF-A- induced monocyte chemotaxis is severely impaired in hypercholesterolemic patients. This reduced response to VEGF seems to be associated with a decreased ability to form functional collaterals.

Therefore we hypothesize that an intensified therapy with atorvastatin 40 mg once a day can significantly improve monocyte function in patients with coronary artery disease and hypercholesterolemia compared to patients who are only treated with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease (angiographically proven)
* diagnosis of hypercholesterolemia (either LDL-C ≥ 4 mmol/l or already treated with lipid-lowering medication)

Exclusion Criteria:

* diabetes mellitus
* uncontrolled arterial hypertension (repeated BP ≥ 160/90 mmHg)
* smoking
* active infections
* acute coronary syndrome (< 8 weeks)
* malignant diseases
* nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-05; Study Completion 2006-03

PRIMARY OUTCOMES:
VEGF-A induced monocyte chemotaxis after 1-month treatment with atorvastatin 40 mg or a placebo once a day
PlGF-1 induced monocyte chemotaxis after 1-month treatment with atorvastatin 40 mg or a placebo once a day
HGF-induced monocyte chemotaxis after 1-month treatment with atorvastatin 40 mg or a placebo once a day
MCP-1-induced monocyte chemotaxis after 1-month treatment with atorvastatin 40 mg or a placebo once a day
VEGF-A+MCP-1-induced monocyte chemotaxis after 1-month treatment with atorvastatin 40 mg or a placebo once a day

SECONDARY OUTCOMES:
HGF+MCP-1-induced monocyte chemotaxis after 1-month treatment with atorvastatin 40 mg or a placebo once a day

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Waltenberger, MD PhD, Principal Investigator — University of Ulm, Germay
Locations (1):
- University Hospital Ulm, Ulm, Germany

REFERENCES:
- [Background] Waltenberger J, Lange J, Kranz A. Vascular endothelial growth factor-A-induced chemotaxis of monocytes is attenuated in patients with diabetes mellitus: A potential predictor for the individual capacity to develop collaterals. Circulation. 2000 Jul 11;102(2):185-90. doi: 10.1161/01.cir.102.2.185. PMID 10889129